CLINICAL TRIAL: NCT02960165
Title: Functional Performance Comparison Between Real and Virtual Tasks in Older Adults
Brief Title: Real and Virtual Tasks in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 39396814.9.1001.0082
Record Dates: First submitted 2016-11-02; First posted 2016-11-09 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Aged

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Virtual interface group A (Experimental): Older adults that started the practice on the virtual interface
  Interventions: Behavioral: Virtual interface group
- Virtual interface group B (Experimental): Older adults that started the practice on the virtual interface and then practiced on real task.
  Interventions: Behavioral: Virtual interface group
- Real interface group A (Active Comparator): Older adults that started the practice on the virtual interface
  Interventions: Behavioral: Real interface group
- Real interface group B (Active Comparator): Older adults that started the practice on the real interface and then practiced on virtual task.
  Interventions: Behavioral: Real interface group

INTERVENTIONS:
Behavioral: Virtual interface group — First practice on virtual interface in order to evaluate the improvement and its influence on real interface performance (second practice).
  Arms: Virtual interface group A; Virtual interface group B
Behavioral: Real interface group — First practice on real interface in order to evaluate the improvement and its influence on virtual interface performance (second practice).
  Arms: Real interface group A; Real interface group B

SUMMARY:
Objective: Evaluate whether a task practiced in virtual environment could provide better performance than the same task in real environment and if performing a task in virtual environment could enable transfer to the same task in real environment and vice versa. Method: the investigators evaluated 65 older adults of both genders, aged 60-82 years. The investigators applied a timing coincident task to measure the perceptual-motor ability to perform a motor response. The participants were divided into two groups: a) started in a real interface and b) started in a virtual interface.

DETAILED DESCRIPTION:
Sixty-five older adults of both sexes (12 males and 53 females) aged 60-82 years (definition used by World Health Organization) were included for participation in the study. Other inclusion criteria included healthy cognitive and motor conditions to understand and perform the required activity, which consisted of scoring more than 24 points on a Mini Mental State Examination administered before testing.

Material and apparatus

The investigators applied the timing coincident task to measure the perceptual-motor ability to perform a motor response in sync with the arrival of an external object at a certain point. This instrument has been widely investigated, especially in the motor learning area. To evaluate the motor learning of the participants using a timing coincident task, two distinct interfaces were applied as follows:

1. Real environment interface (RI): Bassin Anticipation Timer Model 35580 (Lafayette Instrument, Indiana, USA) was used to represent the real environment. This equipment was developed to test the area of visual acuity related to eye-hand coordination and anticipation. The participant was instructed to watch a light as it travels down the runway with 32 LEDs (two runways with 16 red LEDs on each). A cue yellow LED was lit for 0.5 seconds after initiating a test and before the lights run down the runway. The participant must anticipate the light reaching the target (last LED) and press a button to coincide with the arrival of the light at the target. The LCD readout displays the time difference between the response and the arrival of the light at the target and indicate if the response was early or late.
2. Virtual environment interface (VI): The investigators used a virtual coincidence timing task based on the Bassin Anticipation Timer developed by the Department of Electronic Engineering Polytechnic School of the University of São Paulo , and updated by the Information Systems Laboratory of the University of São Paulo. In VI, 10 bubbles represented by 3D design on the computer are displayed simultaneously in a vertical column. The bubble lights change from gray to red sequentially (i.e. from the top to the bottom) until the target and last bubble (the tenth bubble). The task consists of a movement of the hand in a virtual environment produced by the Microsoft Kinect® sensor at the moment the light reaches the target bubble, as proposed in RI task.

Procedure and design The participants were divided into two groups: one group started in RI (RI-group), and the other started in VI (VI-group). Each participant used the dominant hand to perform the tasks (all right-handed). The task was performed in 20 trials for acquisition, 5 trials for retention and 5 trials for transfer. Acquisition and retention were performed at the same velocity, and transfer with an increase of velocity. Both groups performed the tasks in the two interfaces.

The researches provided verbal explanation about the use of instruments before the participants started the tasks. The tasks according to the interfaces are described below.

Virtual interface: Participants were seated on a chair in front of a computer (MS Windows 64bits, Intel® Core™ i7-4810MQ CPU @ 2.80GHz) and Kinect sensor V1.0 to facilitate and enable the task. The image of participant was shown at the top righ of the monitor, and their hand movement in the main screen. The movement to reach the bubble was obtained by Kinect sensor. The participant had to move his/her hand to pass over the target bubble. During acquisition and retention trials, the bubbles simulated a dropped light movement with the turning on and off of the lights in an interval of 500ms (level 4) between position changes, while during transfer light movement was increased with 250ms (level 5) between positions.

Real interface: Participants were standing in front of the Bassin Anticipatory Timer positioned vertically on a table. The standing position was used in the real task to facilitate the participant to be able to see the task with comfort. Participant was orientated that they should press the button when the target light was turned on (synchronously with the target light). The dropped light movement, with the turning on and off of the LEDs occurred at an interval of 100ms (l MPH) between position changes to acquisition and retention phases, and at an interval of 9ms (11MPH) to transfer.

Due to the difference in number of LEDs (RI) and bubbles (VI) between the tasks, to equalize the protocol, the time between the start and end of the task was the same for all phases of the study, i.e., 5 seconds for acquisition and retention and 2.5 seconds for transfer.

ELIGIBILITY:
Inclusion Criteria:

* healthy cognitive and motor conditions to understand and perform the required activity

Exclusion Criteria:

* less than 23 points on a Mini Mental State Examination administered before testing

Ages: 60 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Improvement and transfer of performance through virtual and real task, by using motor learning protocol (acquisition phase, retention and transfer tests) - with one outcome: motor learning. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- School of Arts, Sciences and Humanities of the University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No